CLINICAL TRIAL: NCT04116060
Title: Impact of Dietary Nitrate on Erectile Dysfunction
Brief Title: Dietary Nitrate and Erectile Dysfunction
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Essen (Other)
Responsible Party: Principal Investigator, Fadi Al-Rashid, MD, Principal Investigator, University Hospital, Essen
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: Nitrate E.D.
Record Dates: First submitted 2019-10-03; First posted 2019-10-04 (Actual); Last update posted 2021-01-25 (Actual); Status verified 2021-01

CONDITIONS: Erectile Dysfunction
MeSH Terms: conditions — Erectile Dysfunction

STUDY DESIGN:
Intervention Model Description: Parallel Assignment to intervention vs. control
Who Masked: Participant, Investigator
Masking Description: Double blinded and randomised
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nitrate (Experimental): Dietary nitrate dissolved in water (0,12 mmol sodium-nitrate/kgBW/day) Dietary Supplement: Dietary nitrate 200 ml tab water with 0,12 mmol/kgBW sodium-nitrate
  Interventions: Dietary Supplement: Dietary Nitrate
- Control (Placebo Comparator): Dietary sodium-chloride dissolved in water (0,12 mmol sodium-chloride/kgBW/day) Dietary Supplement: Dietary sodium-chloride 200 ml tab water with 0,12 mmol/kgBW sodium-chloride
  Interventions: Dietary Supplement: Control

INTERVENTIONS:
Dietary Supplement: Dietary Nitrate — Oral dietary nitrate supplementation with (0,12 mmol/kgBW sodium-nitrate)
  Arms: Nitrate
Dietary Supplement: Control — Placebo Comparator: Dietary sodium-chloride dissolved in water (0,12 mmol sodium-chloride/kgBW/day)
  Arms: Control

SUMMARY:
An expanding number of studies suggest a therapeutic role for nitrate and nitrite, most notably in treatment and prevention of cardiovascular disease including ischemia-reperfusion injury and hypertension. The nutritional aspects of these cardioprotective effects are particularly intriguing since nitrate is abundant in our everyday diet. Nitrate improves vascular functions in old adults and improves ischemia reperfusion injury in experimental models.

Whether dietary nitrate improves erectile dysfunction is not known and will be investigated in the present study.

ELIGIBILITY:
Inclusion Criteria:

Patients with erectile Dysfunction (IIEF5: 8-21) PDE-5 Inhibitors Responder Aged 30-80 years

Exclusion Criteria:

* Spinal cord disease
* Insulin dependent Diabetes mellitus
* Prostate cancer after operation, radiotherapy and hormone therapy
* Treatment with NO-Donators or sGC-Activators
* Chronic kidney disease (Stage IV-V)
* Advanced liver dysfunction

Ages: 30 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2020-02-17 (Actual); Primary Completion 2021-06-01 (Estimated); Study Completion 2021-08-01 (Estimated)

PRIMARY OUTCOMES:
The changes of erectile function according to the international index of erectile function (IIEF5) score | 4 Weeks
  Erectile dysfunction improvement as measured by IIEF5 score (range 5-25)

SECONDARY OUTCOMES:
Change in oral microbiome | 4 Weeks
  Change in oral microbiome after dietary nitrate ingestion
Change in cardiac diastolic function, | 4 weeks
  Change in cardiac diastolic function as determined by echocardiography via measurement of E/A and E/e' aggregated to display diastolic function

CONTACTS AND LOCATIONS:
Overall Officials: Tienush Rassaf, Prof, Study Director — University Hospital, Essen; Christos Rammos, MD, Principal Investigator — University Hospital, Essen
Locations (1):
- University Hospital Essen, Essen, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: Undecided